CLINICAL TRIAL: NCT06242496
Title: Brain Abscesses in Transplant Recipients: a Multicentre Retrospective Study
Brief Title: Brain Abscesses in Transplant Recipients: a Multicentre Retrospective Study (BAT-STUDY)
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Sponsor
Other Study IDs: APHP231787
Record Dates: First submitted 2024-01-29; First posted 2024-02-05 (Actual); Last update posted 2024-02-05 (Actual); Status verified 2024-01

CONDITIONS: Brain Abscess
Keywords: Brain abscess; Solid Organ Transplantation; Allogeneic hematopoietic stem cell transplantation; Immunosuppression; Opportunistic infections
MeSH Terms: conditions — Brain Abscess; Opportunistic Infections

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patients with brain abscesses after transplantation
  Interventions: Other: Retrospective follow-up

INTERVENTIONS:
Other: Retrospective follow-up — Data collection

SUMMARY:
Allotransplantation is the process of transferring organ(s), tissue(s) or cell(s) from a healthy donor to a recipient. The two main applications of allotransplantation are solid organ transplantation and allogeneic hematopoietic stem cell transplantation. For several reasons, including the need to use immunosuppressive drugs after transplantation, recipients of allografts carry a high risk of infectious complications.

Central nervous system infections are dreadful complications of transplantation, which can be divided into brain abscesses, meningitis, and encephalitis. In particular, brain abscesses pose major diagnostic and therapeutic challenges to transplant physicians, and are frequently fatal in transplant recipients. As compared with immunocompetent patients, transplant recipients and other immunocompromised patients have an increased risk of brain abscesses due to opportunistic pathogens, including fungi, parasites, bacteria, and mycobacteria.

Determining the epidemiology of brain abscesses is critical to guide transplant teams regarding the diagnosis and management of brain abscesses in transplant recipients.

Because the incidence of brain abscesses is low after transplantation, transplant teams often have limited clinical experience in the management of these infections. Similarly, most publications focusing on post-transplant brain abscesses are either case reports, small case series, or review articles.

We therefore aim to conduct a multicentre retrospective study on the epidemiology, the characteristics, and the outcome of brain abscesses in transplant recipients in the era of new diagnostic tools and progress in prophylaxis.

ELIGIBILITY:
Inclusion Criteria:

* Transplant recipient (i.e., solid organ transplant recipient or allogeneic hematopoietic stem cell transplant recipient)
* Radiological evidence of brain abscess(es) after transplantation
* Brain abscess(es) classified as either proven, probable or possible (see definitions below)Diagnosis of brain abscess made between January 2010 and December 2021

Exclusion Criteria:

* Opposition of the research
* Patients under guardianship

Ages: 0 Years to 100 Years | Sex: All
Age Groups: Child, Adult, Older Adult
Study Population: Patients with brain abscesses after transplantation
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2024-02-01 (Estimated); Primary Completion 2025-02-01 (Estimated); Study Completion 2025-02-01 (Estimated)

PRIMARY OUTCOMES:
Description of the current epidemiology of brain abscesses in transplant recipients | 1 year after brain abscess diagnosis
  Clinical and microbiological characteristics

SECONDARY OUTCOMES:
Comparison of the clinical and microbiological characteristics of brain abscesses between solid organ transplant recipients and allogeneic hematopoietic stem cell transplant recipients | 1 year after brain abscess diagnosis
Compare the clinical and microbiological characteristics of brain abscesses occurring early after transplantation (<M6) with those of brain abscesses occurring later after transplant (> M6) | 1 year after brain abscess diagnosis
Identification of clinical predictors associated with fungal brain abscesses versus brain abscesses due to non-fungal organisms | 1 year after brain abscess diagnosis
Description of the current management of post-transplant brain abscesses in transplant recipients | 1 year after brain abscess diagnosis
  in terms of antimicrobial therapy, immunomodulation, and neurosurgical management
Assessment of the outcome of transplant recipients with brain abscesses | 1 year after brain abscess diagnosis
  i.e. one-year all cause mortality
Identification of factors associated with patient survival in transplant recipients with brain abscesses | 1 year after brain abscess diagnosis

IPD SHARING:
Plan to Share IPD: Undecided